CLINICAL TRIAL: NCT01067638
Title: The Effect of Tranexamic Acid on Postoperative Blood Loss and Coagulation in Patients With Preoperative Anemia Undergoing Off-Pump Coronary Artery Bypass Graft; Double Blind Randomized Control Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Kwak, Young-Lan, Severance Hospital, Dept. of Anesthesiology & Pain Medicine
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2009-0488
Record Dates: First submitted 2010-01-15; First posted 2010-02-11 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Coronary Artery Occlusive Disease
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tranexamic acid (Experimental): Tranexamic Acid on Postoperative Blood loss and Coagulation in Patients with Preoperative Anemia Undergoing Off-Pump Coronary Artery Bypass Graft
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 1.0g loading dose before skin incision and continuous infusion 200 mg/h during surgery

SUMMARY:
The Effect of Tranexamic Acid on Postoperative Blood loss and Coagulation in Patients with Preoperative Anemia Undergoing Off-Pump Coronary Artery Bypass Graft; double blind randomized control study.

ELIGIBILITY:
Inclusion Criteria:

* Fifty patients undergoing OPCAB with preoperative hematocrit levels lower than 35%

Exclusion Criteria:

Patient who has

* Open heart surgery history before
* Thrombosis history
* Myocardial infarction (MI) within 7days recently
* Liver or Kidney disease
* been scheduled emergency surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Tranexamic acid significantly reduce the amount and incidence of homologous transfusion in anemic patients undergoing off-pump coronary artery bypass (OPCAB) | Check the amount 3 times before sugery and 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Univ., Seoul, South Korea